CLINICAL TRIAL: NCT03726346
Title: The Evaluation of the Toffee Mask for the Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA 243
Record Dates: First submitted 2018-10-28; First posted 2018-10-31 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Toffee Full Face Mask (Experimental): Participants will be placed on this arm for a total of 14+- 4 days from visit 2. Participants will be using the Toffee mask during this treatment arm.
  Interventions: Device: Toffee Full Face Mask

INTERVENTIONS:
Device: Toffee Full Face Mask — Participants will be placed on this arm for a total of 14+- 4 days from visit 2. Participants will be using the Toffee mask during this treatment arm.

SUMMARY:
This investigation is a prospective, non-randomized, non-blinded study. This investigation is designed to evaluate the performance, comfort and ease of use of the F&P Toffee mask amongst Obstructive Sleep Apnea (OSA) patients. Up to 45 OSA patients will be recruited from the Pulmonary Disease Specialists Research database.

DETAILED DESCRIPTION:
Visit 1 will involve the participants being consented into the trial. Visit 2 will involve the participants being fitted with the F&P Toffee mask for use in home. The participant will then come in to return the mask (Visit Three) and have a final interview, this ensures the maximum time participants will be exposed to the Toffee mask in home will be 14 ± 4 days from visit two. The mask will be returned to the Institution at the conclusion of the trial and the participant will return to their previous mask. The Institution will recruit all patients within 2 weeks of the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (22+ years of age)
* Able to give informed consent
* Apnea hypopnea Index (AHI) ≥ 5 on diagnostic night
* Either prescribed Automatic positive airway pressure (APAP), Continuous positive airway pressure (CPAP) or Bi-level positive airway pressure (PAP) for OSA
* Fluent in spoken and written English
* Existing OSA mask user

Exclusion Criteria:

* Inability to give informed consent
* Participant intolerant to PAP
* Anatomical or physiological conditions making PAP therapy inappropriate
* Current diagnosis of respiratory disease or carbon Dioxide (CO2) retention
* Pregnant or may think they are pregnant.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Goodwin, Study Director — Research Director; Thomas O'Brien, MD, Principal Investigator — Pulmonologist
Locations (1):
- Pulmonary Disease Specialists, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Toffee Full Face Mask
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Toffee Full Face Mask
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Toffee Mask Acceptability
Description: Participant preference for the Toffee mask over their usual mask. Determined from questionnaires -Subjective
Time Frame: 14±4 days in home
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Full Face Mask
Number analyzed (Participants) | 39
Participants
  Preferred Toffee mask | 27
  Preferred usual mask | 12

2. Primary Outcome: Toffee Mask Comfort
Description: Overall Toffee mask comfort determined from questionnaires-Subjective
Time Frame: 14±4 days in home
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Full Face Mask
Number analyzed (Participants) | 39
Participants
  Very comfortable | 15
  Comfortable | 17
  Neither comfortable nor uncomfortable | 3
  Uncomfortable | 4
  Very uncomfortable | 0

3. Primary Outcome: Toffee Mask Treatment Seal Performance-Subjective
Description: Sealing performance of Toffee mask determined from questionnaires - Subjective
Time Frame: 14±4 days in home
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Full Face Mask
Number analyzed (Participants) | 39
Participants
  Very good | 14
  Good | 14
  Neither good nor poor | 9
  Poor | 2
  Very poor | 0

4. Secondary Outcome: Toffee Mask Treatment Performance-Objective
Description: Objective Apnea Hypopnea Index (AHI) data recorded from the participants Positive Airway Pressure (PAP) device and compared to baseline AHI data - Objective
Time Frame: 14±4 days in home
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Full Face Mask
Number analyzed (Participants) | 39
Participants
  AHI decreased | 19
  AHI increased | 10
  N/A | 10

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for all participants for 1 year from the date informed consent was obtained.
Arm/Group | Toffee Full Face Mask
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 4/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toffee Full Face Mask (N=39)
Cheek pressure/ discomfort (Skin and subcutaneous tissue disorders) | 4 (4) — Cheek pressure/ discomfort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT03726346/Prot_SAP_001.pdf